CLINICAL TRIAL: NCT03922997
Title: An Open-Label, Singe Arm, Multicenter Study to Investigate the Safety and Efficacy of Atezolizumab (Tecentriq) in Previously-Treated Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Investigate the Safety and Efficacy of Atezolizumab in Previously-Treated Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40471
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Participants will receive atezolizumab intravenously on the first day of each cycle. Atezolizumab treatment will continue until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or patient decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1200 mg intravenously on the first day of each 21-day cycle.
  Other Names: Tecentriq

SUMMARY:
This is a phase III, single-arm, multicenter study of the long-term safety and efficacy of atezolizumab treatment in patients with Stage IIIb or Stage IV non-small cell lung cancer (NSCLC) who have progressed following standard systemic chemotherapy (including if given in combination with anti-PD-1 therapy or after anti-PD-1 as monotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Stage IIIb or Stage IV NSCLC that has progressed following standard systemic chemotherapy (including if given in combination with anti-PD-1 therapy or after anti-PD-1 as monotherapy). Patients with a previously detected EGFR mutation or ALK fusion oncogene will be excluded from this study. Overall, patients should not have received more than two lines of systemic chemotherapy. Patients who have discontinued first-line or second-line systemic chemotherapy, targeted therapy, or anti-PD-1 therapy due to intolerance are also eligible.
* The last dose of prior systemic anticancer therapy must have been administered ≥ 21 days prior to the first study treatment.
* The last dose of prior anti-PD-1 therapy must have been administered
* Measurable disease, as defined by Response Evaluation Criteria for Solid Tumors, Version 1.1 (RECIST v1.1)
* Patients with asymptomatic CNS metastases (treated or untreated), as determined by CT or MRI evaluation during screening and prior radiographic evaluation, are eligible
* ECOG performance status 0, 1, or 2
* Life expectancy ≥ 12 weeks
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab
* Patients must have recovered from all acute toxicities from previous therapy, excluding alopecia and toxicities related to prior anti-PD-1-therapy

Exclusion Criteria:

* Patients with EGFR mutation or ALK fusion oncogene
* Symptomatic CNS metastases
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to the first study treatment
* Leptomeningeal disease
* Uncontrolled pericardial effusion or ascites requiring recurrent drainage procedures
* Pregnant or lactating, or intending to become pregnant during the study
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, including significant liver disease
* Significant cardiovascular disease
* Significant renal disorder requiring dialysis or indication for renal transplant
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to study treatment initiation
* Major surgical procedure within 4 weeks prior to study treatment initiation or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
* Prior allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Event Incidence Rates | Baseline up to approximately 3 years
  The incidence of serious adverse events (SAEs) related to atezolizumab.

SECONDARY OUTCOMES:
Overall Survival (OS) Rate | Baseline to 2 years
  Overall survival (OS) rate at 2 years, defined as the proportion of patients remaining alive 2 years after initiation of study treatment
OS | Baseline up to approximately 3 years
  Overall survival (OS), defined as the time from initiation of study treatment to death from any cause
Progression-Free Survival (PFS) | Baseline up to approximately 3 years
  Progression-free survival (PFS), defined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first.
Objective Response Rate (ORR) | Baseline up to approximately 3 years
  Objective response rate (ORR), defined as the percentage of patients who attain complete response (CR) or partial response (PR) according to RECIST v1.1 and also by disease status evaluated by the investigator according to modified RECIST
Duration of Response (DOR) | Baseline up to approximately 3 years
  Duration of response (DOR), defined as the time from initial response to disease progression or death among patients who have experienced a CR or PR (unconfirmed) during the study.
EQ-5D-5L Index-Based and VAS scores | Day 1 of first 3 cycles, then with tumor assessments every 6 weeks for 48 weeks from study treatment date; thereafter every 9 weeks until progressive disease or until treatment discontinuation (up to approximately 3 years)
  EQ-5D-5L, EuroQol 5-Dimension Questionnaire is a self-report health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. The EuroQol EQ-5D has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort and anxiety/depression, as well as a visual analog scale (VAS) that measures health state. Overall scores range from 0 to 1, with low scores representing a higher level of dysfunction.
EORTC QLQ-LC13 score | Day 1 of first 3 cycles, then with tumor assessments every 6 weeks for 48 weeks from study treatment date; thereafter every 9 weeks until progressive disease or until treatment discontinuation (up to approximately 3 years)
  EORTC QLQ-LC13, European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire-Supplemental Lung Cancer Module will be used to assess self-reported outcomes. EORTC QLQ-LC13 includes 13 items that address key lung cancer symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related adverse effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication. The dysphagia scale is multi-item, while the rest are single-item scales.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing
  - Sichuan Cancer Hospital, Chengdu
  - Zhejiang Cancer Hospital; Zhejiang Cancer Hospital cancer department, Hangzhou
  - Harbin Medical University Tumor Hospital; Department of Surgery; Pharmacy, Harbin
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Fudan University Shanghai Cancer Center; Medical Oncology, Shanghai
  - Cancer Hospital Affliated to Xinjiang Medical University, Ürümqi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).